CLINICAL TRIAL: NCT02350660
Title: Oral Immunotherapy for Peanut and Mammalian Meat Allergies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Scott Commins, MD, Associate Professor, Department of Medicine, Allergy and Immunology, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15098
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Food Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cow's milk for alpha-gal allergics (Experimental): daily consumption of cow's milk
  Interventions: Dietary Supplement: cow's milk
- Peanut powder (Experimental): peanut oral immunotherapy
  Interventions: Dietary Supplement: peanut powder

INTERVENTIONS:
Dietary Supplement: cow's milk — daily consumption of cow's milk
  Arms: Cow's milk for alpha-gal allergics
Dietary Supplement: peanut powder — peanut oral immunotherapy
  Arms: Peanut powder

SUMMARY:
Pilot study to assess the effect of oral immunotherapy on specific Immunoglobulin E (IgE) levels and antigen consumption in two distinct food allergies.

DETAILED DESCRIPTION:
In subjects with mammalian meat allergy, the effect of daily oral cow's milk on immune parameters and desensitization will be assessed. Similarly, in subjects with a peanut allergy the effects of low dose peanut flour will be assessed and comparisons between two distinct food allergies.

ELIGIBILITY:
Inclusion Criteria:

* Presence or absence of specific IgE to alpha-gal or peanut

Exclusion Criteria:

* History of severe anaphylaxis
* allergy to cow's milk protein

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Commins, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Wisniewski JA, Commins SP, Agrawal R, Hulse KE, Yu MD, Cronin J, Heymann PW, Pomes A, Platts-Mills TA, Workman L, Woodfolk JA. Analysis of cytokine production by peanut-reactive T cells identifies residual Th2 effectors in highly allergic children who received peanut oral immunotherapy. Clin Exp Allergy. 2015 Jul;45(7):1201-13. doi: 10.1111/cea.12537. PMID 25823600

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to changes in funding structure, the study was unable to be completed with the designed number of participants and was therefore closed to enrollment
Period: Overall Study
Arm/Group | Cow's Milk for Alpha-gal Allergics | Peanut Powder
Started | 7 | 17
Completed | 7 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cow's Milk for Alpha-gal Allergics | Peanut Powder | Total
Number analyzed (Participants) | 7 | 17 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 16 | 16
  Between 18 and 65 years | 6 | 1 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 55 (7) | 8 (3) | 23 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 13 | 16
Region of Enrollment [Number; unit: participants]
  United States | 7 | 17 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Level of Allergen Consumed Post-oral Immunotherapy
Description: consumption of cow's milk or peanut flour at open challenge. This is a single time-point assessment; not measured repeatedly.
Time Frame: Following 36 months of maintenance oral immunotherapy, participants completed an open challenge at month 37
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Cow's Milk for Alpha-gal Allergics | Peanut Powder
Number analyzed (Participants) | 7 | 17
milligrams | 6 (1.3) | 300 (57)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Cow's Milk for Alpha-gal Allergics | Peanut Powder
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/17
Other Adverse Events (participants affected / at risk) | 1/7 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cow's Milk for Alpha-gal Allergics (N=7) | Peanut Powder (N=17)
food intolerance (Gastrointestinal disorders) | 1 (1) | 3 (3) — difficulty tolerating daily dosing

LIMITATIONS AND CAVEATS:
Unblinded and without placebo control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes